CLINICAL TRIAL: NCT05858320
Title: The Impact of an Adaptive Patient-centered Web Application on Medication Optimization in HFrEF Patients (SmartHF)
Brief Title: The Impact of an Adaptive Patient-centered Web Application on Medication Optimization in HFrEF Patients
Acronym: SmartHF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Washington University, Barns Jewish Hospital, St. Louis, MO (Unknown); Henry Ford Hospital, Detroit, MI (Unknown); Emory University, Grady Hospital, Atlanta, GA (Unknown)
Responsible Party: Principal Investigator, Michael Dorsch, Associate Professor of Pharmacy, College of Pharmacy and Clinical Pharmacist, University of Michigan Inpatient Pharmacy Services, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00227631
Record Dates: First submitted 2023-05-01; First posted 2023-05-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SmartHF application (Experimental): The web application-based study intervention provides adaptive medication recommendations that can be shared with their HF provider.
  Interventions: Other: SmartHF application
- Control - Patients Standard Medication(s) (Active Comparator): No change to current medication(s)
  Interventions: Other: SmartHF application

INTERVENTIONS:
Other: SmartHF application — Adaptive medication recommendations that can be shared with the participants HF provider.

SUMMARY:
The SmartHF study is a 12-week prospective randomized controlled multicenter clinical trial. This study will investigate the efficacy of an adaptive web application to facilitate guideline-directed medical therapy (GDMT) optimization in HFrEF patients. Eligible participants will be randomized to the web application intervention or control in a 1:1 manner, stratified by site.

The intervention is an adaptive medication optimization web application that extracts and analyzes the EHR data with a computable medication optimization algorithm. The algorithm provides a medication quality score and outputs medication optimization recommendations written in a patient -friendly manner.

DETAILED DESCRIPTION:
The investigators have developed an adaptive medication optimization web application, named SmartHF, that provides patients with tailored information about potential HFrEF GDMT optimization. SmartHF guides patients to share the GDMT optimization recommendations with their provider during a clinic visit.

Participants will be randomized to receive the web application intervention or control up to 30 days before a clinic visit in a 1:1 manner and followed for 12 weeks after the clinic visit. This trial will determine the efficacy of SmartHF in prescribing GDMT in HFrEF patients compared to controls.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older at screening
2. Diagnosis of heart failure with a left ventricular ejection fraction (LVEF) </= 40% (HFrEF)
3. Have a general medicine provider or general cardiology provider for HFrEF
4. Have internet access and access to their health system's patient portal
5. Fluent in spoken and written English
6. At least two of the following: systolic blood pressure ≥ 110mmg, potassium ≤ 5.5, serum creatinine ≤ 2.5, heart rate ≥ 70
7. At least two eligible heart failure therapies (guideline-recommended BB, RASI, MRA, or SGLT2i) not yet initiated or below 50% of the target dose

Exclusion Criteria:

1. End-stage HF (hospice candidate)
2. Actively treated cancer, except non-melanoma skin cancer
3. Implanted ventricular assist device
4. Current treatment with chronic inotropic therapy
5. Patient's provider for HFrEF care is considered an advanced HF specialist
6. Currently pregnant or intends to become pregnant during the study period
7. Dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint: Change in GDMT medication score | Baseline to Week 12
  Change in GDMT medication score generated by the computable algorithm from baseline to Week 12

SECONDARY OUTCOMES:
Secondary Endpoint: Level of agreement between the medication optimization algorithm recommendations and actual GDMT prescribed | Over 12 Weeks
  The level of agreement between the medication optimization algorithm recommendations (Yes/No) and actual GDMT prescribed (Yes/No)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Emory University, Grady Hospital, Atlanta, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital and Health System, Detroit, Michigan
  - Trinity Healthcare St. Joseph Mercy Ann Arbor, Ypsilanti, Michigan
  - Washington University, Barns Jewish Hospital, St Louis, Missouri

REFERENCES:
- [Background] Dorsch MP, Sifuentes A, Cordwin DJ, Kuo R, Rowell BE, Arzac JJ, DeBacker K, Guidi JL, Hummel SL, Koelling TM. A Computable Algorithm for Medication Optimization in Heart Failure With Reduced Ejection Fraction. JACC Adv. 2023 Apr 12;2(3):100289. doi: 10.1016/j.jacadv.2023.100289. eCollection 2023 May. PMID 38939592